CLINICAL TRIAL: NCT05219461
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Study of the Pharmacokinetics, Safety, and Tolerability of rhEGF Eye Drops in Healthy Male Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability of rhEGF Eye Drops in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: DW_EGF102OP
Record Dates: First submitted 2021-12-29; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A rhEGF 10mcg/mL (Experimental): single dose of rhEGF 10mcg/mL eye drop or single dose of placebo
  *single dose means daily dose (administration twice daily)
  Interventions: Drug: Single dose of rhEGF 10mcg/ml or placebo
- Group B rhEGF 50mcg/mL (Experimental): single dose of rhEGF 50mcg/mL eye drop or single dose of placebo
  *single dose means daily dose (administration twice daily)
  Interventions: Drug: Single dose of rhEGF 50mcg/ml or placebo
- Group C rhEGF 100mcg/mL (Experimental): single dose of rhEGF 100mcg/mL eye drop or single dose of placebo
  *single dose means daily dose (administration twice daily)
  Interventions: Drug: Single dose of rhEGF 100mcg/ml or placebo
- Group D rhEGF 10mcg/mL (Experimental): multiple dose of rhEGF 10mcg/mL eye drop or multiple dose of placebo
  Interventions: Drug: Multiple dose of rhEGF 10mcg/ml or placebo
- Group E rhEGF 50mcg/mL (Experimental): multiple dose of rhEGF 50mcg/mL eye drop or multiple dose of placebo
  Interventions: Drug: Multiple dose of rhEGF 50mcg/ml or placebo
- Group F rhEGF 100mcg/mL (Experimental): multiple dose of rhEGF 100mcg/mL eye drop or multiple dose of placebo
  Interventions: Drug: Multiple dose of rhEGF 100mcg/ml or placebo

INTERVENTIONS:
Drug: Single dose of rhEGF 10mcg/ml or placebo — 6 subjects will be assigned to rhEGF 10mcg/ml eye drop and 2 subjects will be assigned to placebo
  Arms: Group A rhEGF 10mcg/mL
Drug: Single dose of rhEGF 50mcg/ml or placebo — 6 subjects will be assigned to rhEGF 50mcg/ml eye drop and 2 subjects will be assigned to placebo
  Arms: Group B rhEGF 50mcg/mL
Drug: Single dose of rhEGF 100mcg/ml or placebo — 6 subjects will be assigned to rhEGF 100mcg/ml eye drop and 2 subjects will be assigned to placebo
  Arms: Group C rhEGF 100mcg/mL
Drug: Multiple dose of rhEGF 10mcg/ml or placebo — 6 subjects will be assigned to rhEGF 10mcg/ml eye drop and 2 subjects will be assigned to placebo
  Arms: Group D rhEGF 10mcg/mL
Drug: Multiple dose of rhEGF 50mcg/ml or placebo — 6 subjects will be assigned to rhEGF 50mcg/ml eye drop and 2 subjects will be assigned to placebo
  Arms: Group E rhEGF 50mcg/mL
Drug: Multiple dose of rhEGF 100mcg/ml or placebo — 6 subjects will be assigned to rhEGF 100mcg/ml eye drop and 2 subjects will be assigned to placebo
  Arms: Group F rhEGF 100mcg/mL

SUMMARY:
A randomized, double-blind, placebo-controlled, single ascending dose and multiple ascending dose study of the Pharmacokinetics, safety, and tolerability of rhEGF eye drops in healthy male subjects

DETAILED DESCRIPTION:
Primary Objective: To evaluate safety and tolerability of rhEGF eye drop/ Secondary Objective: To evaluate PK of rhEGF eye drop

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged from 20 to 51 at screening test
* Weight 50kg ~100kg BMI 18-27
* Those who are fully understood, voluntarily decided to participate and signed prior to screening
* Those who are deemed suitable for participating in clinical trial due to lab tests, physical exam etc

Exclusion Criteria:

* Those who have clinically significant liver, kidney, respiratory, endocrine, neurologic diseases or hematologic disease, mental diseases(mode disorder, obsessive compulsive disorder)

Ages: 20 Years to 51 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 14 days from baseline
  * sign and symptoms of AE
  * physical exam, vital signs, ECG exam, lab test
  * ophthalmic exam: schirmer's test, TBUT test, slit lamp exam etc
  * Immunogenicity test (anti-drug antibody)

SECONDARY OUTCOMES:
PK characteristics | 14 days from baseline
  Cmax in single dose administration period
PK characteristics | 14 days from baseline
  AUC in single dose administration period
PK characteristics | 14 days from baseline
  Cmax in multiple dose adminitration period
PK characteristics | 14 days from baseline
  AUC in multiple dose administration period
PK characteristics | 14 days from baseline
  Cav in multiple dose administration period

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea